CLINICAL TRIAL: NCT02025153
Title: Comprehensive Pain Programme to Determine Mechanism of Transition of Acute to Chronic Postsurgical Pain- Functional Brain Imaging, Quantitative Sensory Testing, Psychological and Genetic Screening: Prospective Cohort Study
Brief Title: Comprehensive Pain Programme to Determine Mechanism of Transition of Acute to Chronic Postsurgical Pain
Acronym: TAHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/512/D
Record Dates: First submitted 2013-12-29; First posted 2013-12-31 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2017-08

CONDITIONS: Chronic Pain; Anaesthesia; Genetics Predisposition
MeSH Terms: conditions — Chronic Pain; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort (Other): pain testing. All 444 subjects enrolled in the study. Subjects will receive preoperative physical (tonic heat stimulation, mechanical temporal summation and wound hyperalgesia), psychological (State Trait Anxiety Inventory, Pain Catastrophizing Scale), and genetics test; postoperative pain score assessment at 24, 48 hours; postoperative wound hyperalgesia in open abdominal hysterectomy at 72 hours; and phone survey for CPSP at 4 months.
  Interventions: Other: pain testing
- Chronic Post-surgical Pain (Other): pain testing. physical testing, psychological testing, genetics testing and functional brain imaging
  Interventions: Other: pain testing
- No Chronic Post-surgical Pain (Other): pain testing. physical testing, psychological testing, genetics testing and functional brain imaging
  Interventions: Other: pain testing

INTERVENTIONS:
Other: pain testing — physical testing, psychological testing, genetics testing and functional brain imaging

SUMMARY:
To determine whether central sensitization is a mechanism of CPSP (chronic postsurgical pain) in women who will develop CPSP compared to women with no CPSP after hysterectomy. This mechanism is illustrated by a higher pain score in experimental pain models such as tonic heat stimulation, increased evoked mechanical temporal summation and increased wound hyperalgesia.

DETAILED DESCRIPTION:
Chronic pain affects 9% of Singapore population resulting in major socioeconomic burden. Chronic postsurgical pain (CPSP) that persists for over 3 months could be related to nerve injury making this a strategic model to study the transition of acute to chronic pain. CPSP occurs in up to 50% after surgery and up to 32% after hysterectomy. Over 600000 hysterectomies were performed in the US in 2003 making CPSP a significant problem.

Investigators will perform this prospective cohort study to determine whether increased central sensitization and negative psychological experience are involved in the transition of acute to chronic pain after hysterectomy. Investigators will recruit 444 women undergoing hysterectomy and employ validated physical pain testing including tonic heat stimulation, mechanical temporal summation and wound hyperalgesia which had been shown to be related to central sensitization. Pain catastrophizing (negative thoughts of pain) and state trait anxiety scoring will be assessed for the impact of negative cognitive-affective experience on CPSP. A phone survey will be performed at 4 months to determine the primary outcome of CPSP. Arterial spin labeling will be used to delineate cerebral blood flow using arterial spin labeling, functional connectivity and structural connectivity to evaluate insula-anterior cingulate cortex differences in 30 women with CPSP compared to 30 women without CPSP.

In addition to evaluating whether central sensitization, negative psychological experience and activation of brain regions are different in women with CPSP after hysterectomy, the results of this study will elucidate potential mechanisms of CPSP development that will guide in future studies on potential novel therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Anthropometric profile within the following range: age 21-70 yr, American Society of Anesthesiology status I and II women
* Benign condition such as fibroids or adenomyosis
* Abdominal or laparoscopic hysterectomy

Exclusion Criteria:

* Vaginal hysterectomy
* being pelvic pain
* Failure to adequately determine tonic heat stimulation and mechanical temporal summation
* History of drug dependence or recreational drug use
* Allergy to any study drugs

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Chronic postsurgical pain (CPSP) after hysterectomy at 4 months on phone survey | 4 months post hysterectomy
  This is defined as pelvic pain (lower abdominal or perineal pain) in the last week that affected daily living during the 4 months phone survey.
Chronic postsurgical pain (CPSP) after hysterectomy at 6 months on phone survey | 6 months post hysterectomy
  This is defined as pelvic pain (lower abdominal or perineal pain) in the last week that affected daily living during the 6 months phone survey.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | Upon recruitment till 6 months post hysterectomy
  Assessment will be done via Pain Catastrophizing Scale (PCS) questionnaire. Pain catastrophizing refers to the negative thought processes patients have when they are exposed to pain or painful experiences. The PCS is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). It is broken into three subscales being magnification (0-12), rumination (0-16), and helplessness (0-24). A higher value in each subscale indicates a higher tendency to that subscale (worse outcome).
Mechanical Temporal Summation as measured by von Frey filament | 1 day (before surgery)
  Assessment will be done via Mechanical Temporal Summation assessment before surgery. A 180 gram von Frey filament is applied on the subject's forearm. Patient will then be asked to rate the pinprick pain score on a verbal rating scale, 0-100. Following this, 10 consecutive touches at random locations are applied with a 1 second interstimulus interval and within a 1 cm diameter circle. The patient will then be asked to rate the 10th pain score (0-100). The Mechanical Temporal Summation Score is obtained by the difference between the 11th pain score and the 1st pain score. If the score is greater than zero, the patient is implied to have presence of Mechanical Temporal Summation.
State Trait Anxiety Inventory | 1 day
  Assessment will be done via State Trait Anxiety Inventory (STAI) before surgery. STAI is a self-reported tool for assessing anxiety via two sub-scales, each containing 20 items on: i) the state anxiety sub-scale measuring transient anxiety at the time of scoring; and ii) trait anxiety measures dispositional anxiety or anxiety in general.
  Each item in STAI is rated on a 4-point scale: 1 (Not at all) to 4 (very much so). A higher value in each subscale indicates a higher tendency to that subscale (worse outcome on having greater state anxiety or trait anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, Dr, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No